CLINICAL TRIAL: NCT03663270
Title: Influence of the "Hypotension Probability Index" on the Number and Duration of Intraoperative Hypotension in Primary Hip Endoprosthetic Replacement
Brief Title: Hypotension Probability Index in Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Dr. Christian Koch, MD, Principal investigator, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09/17
Record Dates: First submitted 2018-08-28; First posted 2018-09-10 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Hip Disease; Hypotension; Surgery; Anesthesia
Keywords: goal directed management
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Randomized two arm study with two groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Computer generated random list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): HPI monitoring to predict hypotension
  Interventions: Device: Hypotension probability index (HPI)
- Control arm (No Intervention): blinded HPI monitoring

INTERVENTIONS:
Device: Hypotension probability index (HPI) — The intervention group is managed with the HPI parameter to detect and possibly prevent hypotension during anaesthesia.
  Arms: Intervention arm

SUMMARY:
The aim of the study is to investigate the value of the Hypotension Probability Index in reducing intraoperative hypotension in patients with primary hip replacement. The measurement of the blood pressure was and is of great interest for the treating physician/anesthesiologist to optimize the peri- and postoperative patients outcome. The non-invasive measurement can scale the blood pressure but not from heartbeat-to-heartbeat, what results in a loss of information. The invasive measurement by a placed catheter in an artery shows the blood pressure with information about the pulse wave form, the ascending angle, and makes it possible to detect hemodynamic changes in a way the non-invasive blood pressure measurement is lacking. The additional informations of the monitoring and a

DETAILED DESCRIPTION:
Study design The study is designed as a single center randomized prospective interventional trial comparing goal directed hemodynamic management using HPI compared to standard care.

Subcenter University hospital of Giessen, Department of Anesthesiology, Operative Intensive Care and Pain Therapy (Study team: Dres. med. Christian Koch, Emmanuel Schneck, Thomas Zajonz, Dagmar Schulte, Fabian Edinger, Sophie Ruhrmann) 3.3 Study Population The study population is therefore divided into three groups.

1. Intervention group (optimization based on HPI) n=25
2. Control group (optimization based on standard monitoring without HPI) n=25

Inclusion Criteria

* Patients undergoing hip-replacement
* General anesthesia
* Age ≥ 18 years

Exclusion criteria

Predefined exclusion criteria are:

* Participation in another (interventional) study
* Pregnancy and nursing mothers
* Surgery without controlled ventilation
* American Society of Anesthesiologists (ASA) score > III
* Contraindication for invasive blood pressure monitoring
* Renal insufficiency (Kidney Disease Improving Global Outcomes (KDIGO) score Stadium ≥ 2)
* Coagulation disorder

Dropout Criteria None

Patient flow Patients are recruited before surgery after checking inclusion and exclusion criteria. Informed consent is obtained at this time. During this process also basic patients characteristics are obtained:

* Age, sex, height, weight, ASA score
* Pre-existing conditions (hypertension, state after myocardial infarction, coronary heart disease, peripheral arterial disease, renal failure, chronic obstructive pulmonary disease,diabetes)
* Previous surgeries
* Current medication
* Laboratory results

Endpoints

Primary endpoint:

• Frequency (n)/h and Duration (t [min]/% of total anesthesia time) of intraoperative hypotension

Secondary endpoints:

* Suspected reason for hypotension
* Quantity of intravenous volume (crystalloids, colloids, blood products and salvage blood)
* Type and dosage of vasopressors (epinephrine, norepinephrine, dobutamine)
* Cardiac output, cardiac index (CO, CI)
* Stroke volume/ stroke volume index (SV/ SVI)
* Stroke volume variation (SVV)
* Systemic vascular resistance (SVRI)
* Heart rate (HR)
* Blood pressure (BP)
* Duration of surgery, duration of anesthesia
* Blood loss
* Transfusion rate
* Net fluid intake
* Additional outcome parameter

  * hospital length of stay
  * intensive care length of stay
  * duration of mechanical ventilation
  * hemoglobin level at the end of surgery

Data Processing Data collection is carried out consistently on pre-defined time-points in our electronic patient data management system (NarkoData, IMESO Company, Giessen, Germany) into a separated study database(Microsoft Excel). Patient data is transferred to the database as pseudonyms based on a random key method. The chart with the patient data and decrypting keys is kept in the study center for at least 15 years after the end of the study (publication). Data anonymization is intentionally not performed to give patients the option for data insight or deletion of their data in the future.

Data management and evaluation is performed by the study team.

Patient number and Biometrics The aim of the study is to show the benefit of early and automated monitoring of intraoperative hypotension index in order to support automatically registration of the approach of critical situations given as probability of occurrence of hypotension.

Benefit - Risk assessment Potential benefit Based on a continuous monitoring by additional monitoring system (HPI) an early detection of potential life threatening events is possible. This can result in an optimization of the patients' therapy and a better outcome.

Potential Risks The presented study is an interventional study. The potential risks are marginal. The usage of an arterial catheter is based on preexisting diseases, to monitor the blood pressure continuously. The risk of arterial injuries, infection, fistula etc. is minimal. The time points of blood samples for the study are in line with routine sampling. Based on this, there is no additional risk for the patient.

Benefit/ Risk analysis The benefit for the patients is additional monitoring, based on an additional monitoring device and the supervising study doctor, who can support the treating anesthesiologist with information in potentially critical situations. Thereby, it is possible to treat early goal-directed and possibly improve the patients outcome. Considering the potential benefits of the generated information for the patient in comparison to the expected risks, the beneficial effect is overbalanced.

The expected gain in knowledge from this study could be used for optimizing perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip-replacement

  * General anesthesia
  * Age ≥ 18 years

Exclusion Criteria:

* Participation in another (interventional) study

  * Pregnancy and nursing mothers
  * Surgery without controlled ventilation
  * ASA > III
  * Contraindication for invasive blood pressure monitoring
  * Renal insufficiency KDIGO Stadium ≥ 2
  * Coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Episode of hypotension | up to 18 months
  The aim of the study is to investigate whether a goal directed treatment according to the Hypotension Probability Index compared to standard care can reduce the incidence of intraoperative hypotension in patients with hip-replacement. As primary endpoints frequency (n)/h, absolute and relative duration (t [min]/% of total anesthesia time) of intraoperative hypotension were defined for this study.

SECONDARY OUTCOMES:
Changes of fluid management | up to 18 months
  Amount of of intravenous fluids (ml of crystalloids, ml of colloids)
Changes of catecholamine management | up to 18 months
  Dosage of vasopressors and inotropes (µg)

CONTACTS AND LOCATIONS:
Locations (1):
- Michael Sander, Giessen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schneck E, Schulte D, Habig L, Ruhrmann S, Edinger F, Markmann M, Habicher M, Rickert M, Koch C, Sander M. Hypotension Prediction Index based protocolized haemodynamic management reduces the incidence and duration of intraoperative hypotension in primary total hip arthroplasty: a single centre feasibility randomised blinded prospective interventional trial. J Clin Monit Comput. 2020 Dec;34(6):1149-1158. doi: 10.1007/s10877-019-00433-6. Epub 2019 Nov 29. PMID 31784852